CLINICAL TRIAL: NCT04372121
Title: A Double-blind Randomized Extension Study to Assess the Long-term Efficacy and Safety of Linzagolix in Subjects With Endometriosis-associated Pain
Brief Title: Extension to Study on Efficacy and Safety of Linzagolix for the Treatment of Endometriosis-associated Pain
Acronym: EDELWEISS 5
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study is an extension of Study 18-OBE2109-002 that has been terminated due to enrolment challenges. Consequently, this study has also been terminated.
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-OBE2109-005
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2021-12

CONDITIONS: Endometriosis
Keywords: Dysmenorrhea; Dyspareunia; Dyschezia; Non-menstrual pelvic pain
MeSH Terms: conditions — Endometriosis; Dysmenorrhea; Dyspareunia; Constipation | interventions — linzagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Linzagolix 75 mg (Experimental)
  Interventions: Drug: 75 mg linzagolix tablet; Drug: Placebo tablet to match 200 mg linzagolix tablet; Drug: Placebo capsule to match Add-back capsule
- Linzagolix 200 mg + Add-back (E2 1 mg / NETA 0.5 mg) (Experimental)
  Interventions: Drug: 200 mg linzagolix tablet; Drug: Add-back capsule (E2 1 mg / NETA 0.5 mg); Drug: Placebo tablet to match 75 mg linzagolix tablet

INTERVENTIONS:
Drug: 75 mg linzagolix tablet — For oral administration once daily
  Arms: Linzagolix 75 mg
Drug: 200 mg linzagolix tablet — For oral administration once daily
  Arms: Linzagolix 200 mg + Add-back (E2 1 mg / NETA 0.5 mg)
Drug: Add-back capsule (E2 1 mg / NETA 0.5 mg) — For oral administration once daily
  Arms: Linzagolix 200 mg + Add-back (E2 1 mg / NETA 0.5 mg)
Drug: Placebo tablet to match 75 mg linzagolix tablet — For oral administration once daily
  Arms: Linzagolix 200 mg + Add-back (E2 1 mg / NETA 0.5 mg)
Drug: Placebo tablet to match 200 mg linzagolix tablet — For oral administration once daily
  Arms: Linzagolix 75 mg
Drug: Placebo capsule to match Add-back capsule — For oral administration once daily
  Arms: Linzagolix 75 mg

SUMMARY:
The primary objective of this extension study is to assess the maintenance of efficacy of linzagolix administered orally once daily for up to an additional 6 months (for up to 12 months of treatment in total) in women who have already completed 6 months of linzagolix treatment at a dose of 75 mg alone or of 200 mg in combination with ABT (E2 1 mg / NETA 0.5 mg), in the management of moderate to severe endometriosis-associated pain (EAP) in women with surgically confirmed endometriosis.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind study. Subjects who have completed the 6-month Treatment Period in 18-OBE2109-002 - Edelweiss 2 study (herein referred to as main study) will be invited to enter the present extension study. Month 6 visit of the main study is a decision point for Subjects to either end treatment and enter a post-treatment follow up (part of the main study), or to opt for a 6-month treatment extension. All subjects will receive once daily either linzagolix 75 mg alone (with ABT placebo) or 200 mg combined with ABT for 6 months. Subjects who received placebo during the main study will be randomized to either linzagolix 75 mg alone (with ABT placebo) or linzagolix 200 mg with ABT. Subjects who received active treatment during the main study will continue with the same treatment. Double-dummy design will be used in order to maintain the blinding of the study.

After end of treatment in the extension study (6-month treatment period: from Month 6 to Month 12), subjects will enter a post-treatment Follow-Up Period of 6 months with no investigational medicinal product (IMP) or - for subjects willing to continue treatment - a second extension study will be proposed.

ELIGIBILITY:
Inclusion Criteria:

The subject must have:

* completed the 6-month treatment in the main study
* agreed to continue to use only the analgesic rescue medication permitted by the protocol during the Treatment and Follow-up Periods
* agreed to continue to comply with the requirements of the study protocol for the duration of the extension study

Exclusion Criteria:

The subject will be excluded if she:

* is pregnant or breast feeding or is planning a pregnancy within the duration of the of the study (including the Follow-up Period)
* likely to require treatment during the study with any of the restricted medications
* has any other clinically significant gynecologic condition identified during the main study on transvaginal ultrasound (TVUS), on endometrial biopsy or at the manual breast examination, which might interfere with the study efficacy and safety objectives
* meets any of the main study discontinuation criteria

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-02-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (23):
  - Applied Res Center of Ar / Id # 735, Little Rock, Arkansas
  - Futura Research, Inc. / ID # 781, Norwalk, California
  - Adv Womens Health Institute / ID # 761, Greenwood Village, Colorado
  - Red Rocks OB/GYN / ID # 732, Lakewood, Colorado
  - Dr. David I. Lubetkin, LLC / ID # 703, Boca Raton, Florida
  - Coral Way Research / ID # 799, Miami, Florida
  - La Salud Research Clinic, Inc. / ID # 824, Miami, Florida
  - A Premier Medical Research of Florida, LLC / ID # 752, Orange City, Florida
  - Clinical Associates of Orlando, LLC / ID # 779, Orlando, Florida
  - Providea Health Partners LLC / ID # 734, Evergreen Park, Illinois
  - Onyx Clinical Research / ID # 793, Flint, Michigan
  - Valley OBGYN / ID # 704, Saginaw, Michigan
  - ClinOhio Res Services, LLC / ID # 722, Columbus, Ohio
  - Complete Healthcare for Women / ID # 801, Columbus, Ohio
  - Hilltop OBGYN / ID # 711, Franklin, Ohio
  - Clinical Research Associates Inc / ID # 802, Nashville, Tennessee
  - Austin Area ObGyn PLLC / ID # 701, Austin, Texas
  - OB/GYN North Austin / ID # 764, Austin, Texas
  - HCWC dba DiscoveryClinical Trials / ID # 771, Dallas, Texas
  - Signature Gyn Services / ID # 726, Fort Worth, Texas
  - Medical Colleagues of Texas / ID # 819, Katy, Texas
  - Maximos OB/GYN, League City, Texas
  - Physicians Research Options / ID # 766, Draper, Utah
- CARe Clinic / ID # 872, Red Deer, Alberta, Canada
- Puerto Rico Medical Res Inc. / ID # 890, Ponce, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 85 subjects randomized in the Edelweiss 2 study, 37 completed the 6-month treatment. Of the 37 subjects, 30 subjects opted to participate in the current extension study (7 from Placebo, 13 from LGX 75 mg, and 10 from LGX 200 mg+ABT). At entry into the extension study, the 7 subjects in the placebo group were re-randomized to an active LGX group (PBO/LGX 75 mg: 3, PBO/LGX 200 mg+ABT: 4). Subjects receiving LGX during Edelweiss 2 study, continued treatment as randomized in the main study.
Pre-assignment Details: Subjects who received placebo in the main study were randomized in a 1:1 ratio to either linzagolix 75 mg alone (with ABT-matching placebo) or linzagolix 200 mg with ABT, as per the main study randomization schedule.
Groups:
- LGX 75 mg: [Main study: 6 months] The IMPs mentioned below were administered once daily orally.
  * 1 x Linzagolix 75 mg tab.
  * 1 x Linzagolix 200 mg placebo tab.
  * 1 x ABT placebo cap.
  [Extension study: 6 months] Same treatment as the main study
- LGX 200 mg+ABT: [Main study: 6 months] The IMPs mentioned below were administered once daily orally.
  * 1 x Linzagolix 200 mg tab.
  * 1 x Linzagolix 75 mg placebo tab.
  * 1 x ABT cap. (E2 1 mg / NETA 0.5 mg)
  [Extension study: 6 months] Same treatment as the main study
- Placebo/LGX 75 mg: [Main study: 6 months] The IMPs mentioned below were administered once daily orally.
  * 1 x Linzagolix 75 mg placebo tab.
  * 1 x Linzagolix 200 mg placebo tab.
  * 1 x ABT placebo cap.
  [Extension study: 6months] Same treatment as LGX 75 mg group in the extension study
- Placebo/LGX 200 mg+ABT: [Main study: 6 months] The IMPs mentioned below were administered once daily orally.
  * 1 x Linzagolix 75 mg placebo tab.
  * 1 x Linzagolix 200 mg placebo tab.
  * 1 x ABT placebo cap
  [Extension study: 6 months] Same treatment as LGX 200 mg+ABT group in the extension study
Period: Overall Study
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo/LGX 75 mg | Placebo/LGX 200 mg+ABT
Started | 13 | 10 | 3 | 4
Completed | 3 | 4 | 1 | 2
Not Completed | 10 | 6 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0
Not completed — Study termination | 6 | 5 | 1 | 1
Not completed — Hysterectomy planned | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo/LGX 75 mg | Placebo/LGX 200 mg+ABT | Total
Number analyzed (Participants) | 13 | 10 | 3 | 4 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 3 | 4 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.6 (6.0) | 30.6 (7.7) | 29.0 (7.2) | 31.5 (7.1) | 31.9 (6.7)
Age, Customized [Median (Inter-Quartile Range); unit: Years] | 34.0 [29.0 to 36.0] | 30.5 [27.0 to 35.0] | 31.0 [21.0 to 35.0] | 33.5 [26.0 to 37.0] | 32.0 [28.0 to 36.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 3 | 4 | 30
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 1 | 1 | 10
  Not Hispanic or Latino | 10 | 5 | 2 | 3 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 12 | 9 | 3 | 4 | 28
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 1 | 0 | 0 | 1
  Puerto Rico | 2 | 1 | 0 | 0 | 3
  United States | 11 | 8 | 3 | 4 | 26
Weight [Mean (Standard Deviation); unit: kg] | 80.992 (14.425) | 76.446 (22.398) | 72.910 (29.701) | 76.143 (27.300) | 77.979 (18.972)
BMI [Mean (Standard Deviation); unit: kg/m2] | 29.650 (4.27) | 28.390 (9.01) | 28.230 (9.46) | 27.300 (6.86) | 28.770 (6.67)

OUTCOME MEASURES:

1. Primary Outcome: Dysmenorrhea
Description: Monthly Severity Data of dysmenorrhea (DYS) at Month 6 were measured on a 4-point (0: No pain, 1: Mild pain, 2: Moderate pain, 3: Severe pain) Verbal Rating Scale (VRS). The "Mean±SD" of Monthly Severity Data for each treatment arm were calculated and provided as the efficacy data.
Time Frame: 6 Months
Population: Of the 37 subjects who completed the main study (NCT03986944), 30 subjects participated in the extension study (NCT04372121). Of these 30, there were no subjects who had the Monthly Severity Data of DYS and/or NMPP on Day 1 or Month 12 to evaluate the efficacy but there were 5 subjects that had Monthly Severity Data on Month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo/LGX 75 mg | Placebo/LGX 200 mg+ABT
Number analyzed (Participants) | 1 | 1 | 2 | 1
score on a scale | 2.0 (0.0) | 2.0 (0.0) | 2.5 (0.5) | 2.0 (0.0)

2. Primary Outcome: Non-menstrual Pelvic Pain
Description: Monthly Severity Data of non-menstrual pelvic pain (NMPP) at Month 6 were measured on a 4-point (0: No pain, 1: Mild pain, 2: Moderate pain, 3: Severe pain) Verbal Rating Scale (VRS). The "Mean±SD" of Monthly Severity Data for each treatment arm were calculated and provided as the efficacy data.
Time Frame: 6 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo/LGX 75 mg | Placebo/LGX 200 mg+ABT
Number analyzed (Participants) | 1 | 1 | 2 | 1
score on a scale | 1.0 (0.0) | 2.0 (0.0) | 2.5 (0.5) | 2.0 (0.0)

ADVERSE EVENTS:
Time Frame: Month 6 to Month 12 of the treatment period
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical trial subject administered an investigational medicinal product (IMP) and which did not necessarily have a causal relationship with this treatment. Therefore, AE was any unfavourable sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an IMP, whether or not considered related to the IMP.
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo/LGX 75 mg | Placebo/LGX 200 mg+ABT
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/10 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 4/13 | 4/10 | 0/3 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LGX 75 mg (N=13) | LGX 200 mg+ABT (N=10) | Placebo/LGX 75 mg (N=3) | Placebo/LGX 200 mg+ABT (N=4)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LGX 75 mg (N=13) | LGX 200 mg+ABT (N=10) | Placebo/LGX 75 mg (N=3) | Placebo/LGX 200 mg+ABT (N=4)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The main study (NCT03986944) was prematurely terminated by the impact of the COVID-19 pandemic. As a result, the extension study (NCT04372121) was also terminated early before enough subjects could be enrolled and treated for the evaluation of the planned efficacy endpoints. So, we quantified the Monthly Severity Data at Month 6 for the 5 subjects (i.e. 0: No pain, 1: Mild pain, 2: Moderate pain, 3: Severe pain) and showed the "Mean±SD" for each treatment arm as the efficacy data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT04372121/Prot_002.pdf
  • Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT04372121/SAP_003.pdf